CLINICAL TRIAL: NCT01199224
Title: A Phase 1, Single-Dose, Randomized, Group Sequential Cross-Over Study Evaluating the Bioavailability and Food Effect of Three Formulations of Veliparib on Pharmacokinetics in Subjects With Solid Tumors
Brief Title: To Determine the Food Effect and Bioavailability of Three Formulations of Veliparib in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M11-846
Record Dates: First submitted 2010-07-19; First posted 2010-09-10 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2010-12

CONDITIONS: Solid Tumors
Keywords: Solid Tumors; veliparib; refractory; relapsed
MeSH Terms: conditions — Recurrence | interventions — veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Experimental)
  Interventions: Drug: veliparib
- Arm B (Experimental)
  Interventions: Drug: veliparib
- Arm C (Experimental)
  Interventions: Drug: veliparib
- Arm D (Experimental)
  Interventions: Drug: veliparib

INTERVENTIONS:
Drug: veliparib — veliparib formulation A
  Other Names: ABT-888
  Arms: Arm A
Drug: veliparib — veliparib formulation B
  Other Names: ABT-888
  Arms: Arm B
Drug: veliparib — veliparib formulation C
  Other Names: ABT-888
  Arms: Arm C
Drug: veliparib — veliparib formulation C
  Other Names: ABT-888; velaparib
  Arms: Arm D

SUMMARY:
Compare the bioavailability of three veliparib formulations in subjects with solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with cytologically/histologically confirmed solid tumors that are either relapsed or refractory to standard therapy or there is no known effective therapy.
2. In the opinion of the Investigator, life expectancy is 12 weeks or greater.
3. Subjects with known brain metastases must have clinically controlled neurologic symptoms, defined as surgical excision and/or radiation therapy followed by 21 days of stable neurologic function and no evidence of central nervous system (CNS) disease progression as determined by computed tomography (CT) scan or magnetic resonance imaging (MRI) within 21 days prior to the first dose of study drug.
4. Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 2.
5. Subject must have adequate bone marrow, renal and hepatic function per local laboratory reference range.

Exclusion Criteria:

1. The subject is unable to swallow capsules or has nausea or vomiting.
2. Female subject is pregnant or breast-feeding.
3. Subject has a history of or an active medical condition(s) that affects absorption or motility (e.g., Crohn's disease, celiac disease, gastroparesis, short bowel syndrome).
4. History of gastric surgery, vagotomy, bowel resection (except for left hemicolectomy) or any surgical procedure that might interfere with gastrointestinal motility, potentiometric hydrogen ion concentration (pH) or absorption.
5. Subject exhibits evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

   * Known seizure disorder that is uncontrolled over the past month
   * Active uncontrolled infection
   * Unstable angina pectoris or cardiac arrhythmia
   * Psychiatric illness/social situation that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Assess the oral bioavailability of veliparib | Up to 4 weeks.
  Assess the relative bioavailability of Formulation A, Formulation B and Formulation C with or without food measured using area under the plasma concentration-time curve (AUC), the maximum observed plasma concentration (Cmax), and time to Cmax (Tmax).

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of veliparib in patients with solid tumors | Up to 4 weeks
  Safety and tolerability will be assessed through clinical laboratory tests, electrocardiograms (ECGs), vital signs, physical exams and adverse event assessments

CONTACTS AND LOCATIONS:
Overall Officials: Bhardwaj Desai, MD, Study Director — Abbott

REFERENCES:
- [Result] Mostafa NM, Chiu YL, Rosen LS, Bessudo A, Kovacs X, Giranda VL. A phase 1 study to evaluate effect of food on veliparib pharmacokinetics and relative bioavailability in subjects with solid tumors. Cancer Chemother Pharmacol. 2014 Sep;74(3):583-91. doi: 10.1007/s00280-014-2529-2. Epub 2014 Jul 23. PMID 25053388